CLINICAL TRIAL: NCT04801758
Title: Antiretroviral Analytical Treatment Interruption (ATI) to Assess Immunologic and Virologic Responses in Participants Who Received VRC01 or Placebo and Became HIV-infected During HVTN 704/HPTN 085
Brief Title: Analytical Treatment Interruption (ATI) to Assess the Immune System's Ability to Control HIV in Participants Who Became HIV-infected During the HVTN 704/HPTN 085 AMP Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HIV Vaccine Trials Network (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); HIV Prevention Trials Network (Network); Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HVTN 804/HPTN 095; UM1AI068614 (NIH)
Record Dates: First submitted 2021-03-01; First posted 2021-03-17 (Actual); Results first posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: HIV Infection
Keywords: HIV; Antibody; LTNPs; ECs; VCs; Treatment interruption
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Analytical Treatment Interruption (Experimental): Participants who received VRC01 or placebo and got HIV while enrolled in HVTN 704/HPTN 085 (NCT02716675).
  Interventions: Other: Analytical Treatment Interruption

INTERVENTIONS:
Other: Analytical Treatment Interruption — Participants will stop taking their HIV medication and will stay off HIV medication unless and until the HIV levels in their blood show that their immune system is not controlling their HIV or they meet other ART re-start criteria as noted in section "Detailed Description".

SUMMARY:
The purpose of this study is to learn whether having the AMP Study antibody (called VRC01) in a person's body might help their immune system control HIV better, even without HIV medication called antiretroviral therapy or ART, if they get HIV. This study will evaluate the viral and immune system responses in an Analytical Treatment Interruption (ATI), in participants who received VRC01 or placebo and got HIV while enrolled in HVTN 704/HPTN 085 (NCT02716675).

Participants in this study will stop taking their HIV medication. They will stay off HIV medication unless and until the HIV levels in their blood show that their immune system is unable to control the HIV or they meet other ART re-start criteria as noted in section "Detailed Description". While they are not taking HIV medication, their HIV levels will be tested frequently, and their health will be monitored closely. This is called an analytical treatment interruption, or an ATI. An ATI is an experimental procedure that is only used in carefully monitored research.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate immunologic and virologic responses in an Analytical Treatment Interruption (ATI), in participants who received VRC01 or placebo and got HIV while enrolled in the HVTN 704/HPTN 085 Antibody-Mediated Prevention (AMP) Study (NCT02716675).

ATI begins with the cessation of ART on Schedule 1 (Monitoring ATI). Participants on Schedule 1 will attend study visits every week for the first 8 weeks and at least every 2 weeks for the next 16 weeks. After that, participants will attend study visits once a month for the next 6 months, if their body is controlling their HIV without ART. Participants on Schedule 1 for more than a year will have visits every 3 months.

For participants on Schedule 1 (Monitoring ATI), a confirmed VL ≥ 200 copies/mL will trigger transition to Schedule 2 (ATI monitoring with viremia). Participants on Schedule 2 will attend study visits every week for the first 8 weeks and at least every 2 weeks for the next 28 weeks. After that, participants will attend study visits once a month for the next 4 months, if their body is controlling their HIV without ART. Participants on Schedule 2 for more than a year will have visits every 3 months.

For participants on Schedule 1 (Monitoring ATI), any of the following non-virologic criteria will trigger re-initiation of ART and transition to Schedule 3 (Follow-up on ART) : confirmed CD4+ T-cell count < 350 cells/mm3, any HIV-related syndrome, pregnancy or breastfeeding, or ART re-initiation requested by participant or if deemed medically necessary by primary HIV provider or clinical research site Investigator of Record. Participants on Schedule 3 will attend study visits every 2 weeks for the first 12 weeks, once a month for the next 16 weeks, and on 2 occasions 3 months apart for the next 24 weeks.

For participants on Schedule 2 (ATI monitoring with viremia), the following virologic criteria will trigger re-initiation of ART and transition to Schedule 3 (Follow-up on ART): viral load remains ≥ 1,000 copies/mL for ≥ 4 consecutive weeks AND viral load has not dropped 0.5 log from the previous week (Week 0 - Week 24), confirmed viral load ≥ 200 copies/mL (after Week 24). Or, the following non-virologic criteria will trigger re-initiation of ART and transition from Schedule 2 (ATI monitoring with viremia) to Schedule 3 (Follow-up on ART): confirmed CD4+ T-cell count < 350 cells/mm3, any HIV-related syndrome, pregnancy or breastfeeding, or ART re-initiation requested by participant or if deemed medically necessary by primary HIV provider or clinical research site Investigator of Record.

Study duration is potentially indefinite for participants maintaining extreme and extended viral control during ATI. Study duration for most participants is expected to be 13-18 months. The maximum anticipated duration for any participant is expected to be approximately 2 1/2 to 3 years.

Visits may include medical history review, physical exam, HIV testing, other STI testing (blood, urine, and rectal and oral swab collection), blood draws, pregnancy testing for participants assigned female sex at birth that can become pregnant, HIV transmission risk reduction counseling, and interviews/questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Estimated date of HIV-1 acquisition within 8 weeks of participant's last HVTN 704/HPTN 085 infusion.
* Initiated ART within 28 weeks of HVTN 704/HPTN 085 HIV-1 date of diagnosis.
* Receiving continuous ART for at least 1 year. ART interruptions of up to 7 days and ≥ 90 days prior to enrollment are acceptable. Within- and between-class changes in ART within the previous year are acceptable.
* If on an NNRTI, willingness and ability to switch to a PI- or INSTI-containing regimen for at least 4 weeks prior to ART interruption.
* Willingness to interrupt ART for up to 24 weeks or up to the time of meeting ART re-initiation criteria.
* Willingness to re-initiate ART upon meeting study ART re-initiation criteria.
* Willingness to use barrier protection (ie, male or female condoms) for all sexual activity until after confirmation of viral suppression following ART re-initiation.
* Willingness for CRS staff to contact primary HIV care provider to exchange information regarding HVTN 804/HPTN 095 and participant medical history.
* Site investigator anticipates that a fully active alternative ART regimen could be constructed and would be available in the event of virologic failure on the participant's current ART regimen.
* Access to a participating CRS and willingness to adhere to study visit schedule and to be followed for the planned duration of the study.
* Ability and willingness to provide informed consent.
* Assessment of understanding: volunteer demonstrates understanding of this study; completes a questionnaire prior to enrollment with verbal demonstration of understanding of all questionnaire items answered incorrectly.
* Agrees not to enroll in another study of an investigational research agent for the duration of the participant's trial participation.

Laboratory Inclusion Values:

Immunology/Virology

* HIV-1 infection, with reactive HIV-1 antibody and any Multispot or Geenius HIV-1/HIV-2 results, documented by the HVTN 704/HPTN 085 HIV diagnostic algorithm.
* Plasma HIV-1 RNA ≥ 1,000 copies/mL by any assay, prior to initiating ART.
* CD4+ cell count ≥ 450 cells/mm3 obtained within 90 days prior to enrollment.
* One plasma HIV-1 RNA below the lower limit of quantitation (LLOQ) of an VQA-certified or DAIDS-approved assay and collected:

  * at screening, within 90 days prior to enrollment; and
  * greater than 9 months prior to the screening HIV-1 RNA.

Hematology

* Hemoglobin (Hgb) ≥ 10.0 g/dL for volunteers who were assigned female sex at birth, ≥ 11.0 g/dL for volunteers who were assigned male sex at birth.
* Absolute neutrophil count (ANC) ≥ 750 cells/mm3
* Platelets ≥ 100,000 cells/mm3

Chemistry

* ALT < 2.5 times the institutional upper limit of normal and direct bilirubin within the institutional range of normal.
* Estimated glomerular filtration rate (eGFR) > 60 mL/min/1.73m2

Reproductive Status

* Volunteers capable of becoming pregnant: negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test performed at the screening visit and prior to enrollment. Persons who are NOT capable of becoming pregnant due to having reached menopause (no menses for 1 year) or having undergone total hysterectomy or bilateral oophorectomy or tubal ligation (verified by medical records) are not required to undergo pregnancy testing.
* Reproductive status: A volunteer who is capable of becoming pregnant must agree to consistently use effective contraception for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment through confirmation of viral suppression following ART re-initiation.
* Volunteers capable of becoming pregnant must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization, until after confirmation of viral suppression following ART re-initiation.

Exclusion Criteria:

1. Any plasma HIV-1 RNA ≥ LLOQ (LLOQ: 75, 50, 40, or 20 copies/mL) within 12 months prior to enrollment.

   • NOTE: Two "blips" (ie, plasma HIV-1 RNA > LLOQ) < 400 copies/mL are allowed if preceded and followed by values < LLOQ and if the blips occur more than 6 months prior to enrollment.

   Note: US volunteers must have results from a CLIA or VQA-approved assay. Non-US sites must have results from locally available assays that are approved as standard-of-care by their regional governing bodies.
2. History of AIDS-defining illnesses or US Centers for Disease Control (CDC) Category C events per the current list on the CDC website (see HVTN 804/HPTN 095 SSP).
3. Autoimmune disease, including Type I diabetes mellitus (Not excluded from participation: Volunteer with mild, stable and uncomplicated autoimmune disease that does not require consistent immunosuppressive medication and that, in the judgment of the site investigator, is likely not subject to exacerbation and likely not to complicate AE assessments).
4. Immunosuppressive medications received within 6 months before enrollment (Not exclusionary: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatologic condition; or [4] a single course of oral/parenteral prednisone or equivalent at doses < 60 mg/day and length of therapy < 11 days with completion at least 30 days prior to enrollment).
5. Blood products received within 120 days before planned ART interruption.
6. Investigational research agents, other than experimental vaccine(s) (See Exclusion Criterion #7), received within 30 days before planned ART interruption.
7. HIV or non-HIV experimental vaccine(s) received within the last 1 year. Exceptions may be made by the HVTN 804/HPTN 095 PSRT for vaccines that have subsequently undergone licensure by the FDA or by the national regulatory authority where the volunteer is enrolling. For volunteers who have received control/placebo in an experimental vaccine trial, the HVTN 804/HPTN 095 PSRT will determine eligibility on a case-by-case basis. For volunteers who have received an experimental vaccine(s) greater than 1 year ago, eligibility for enrollment will be determined by the HVTN 804/HPTN 095 PSRT on a case-by-case basis.
8. Licensed live attenuated vaccines received within 30 days before planned ART interruption (eg, measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever; live attenuated influenza vaccine).
9. Licensed vaccines that are not live attenuated vaccines received within 14 days before planned ART interruption (eg, tetanus, pneumococcal, hepatitis A or B).
10. Receipt of any emergency-use authorized, WHO emergency use listed, licensed or registered SARS-CoV-2 (severe acute respiratory syndrome coronavirus 2) vaccine within 4 weeks before planned ART interruption. Note: SARS-CoV-2 vaccination is not required for HVTN 804/HPTN 095 eligibility.
11. Significant or unstable cardiac or cerebrovascular disease (eg, angina, congestive heart failure [CHF], recent cerebrovascular accident [CVA], or myocardial infarction [MI]).
12. Hepatitis B surface antigen (HBsAg) or positive HCV RNA (Not exclusionary: positive HCV Ab with negative HCV RNA).
13. Volunteers who have:

    * a SARS-CoV-2 positive test (direct viral detection, eg, viral nucleic acid or antigen detection) ≤14 days of enrollment, if asymptomatic OR
    * unresolved COVID-19 (ie, SARS-CoV-2 positive test AND symptoms) ≤ 14 days of enrollment (not excluded: individuals with symptoms consistent with residual sequelae of resolved COVID19, in the clinical judgement of the investigator)
14. Pregnant or breastfeeding
15. Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

    * A process that would affect the immune response;
    * A process that would require medication that affects the immune response;
    * Any contraindication to repeated blood draws, including inability to establish venous access;
    * A condition that requires active medical intervention or monitoring to avert grave danger to the volunteer's health or well-being during the study period; or
    * Any condition specifically mentioned among the exclusion criteria.
16. Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety, or a volunteer's ability to give informed consent.
17. Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, could be exacerbated by events associated with protocol participation, which include: ATI, low-level viremia, subsequent viral rebound, and ART re-initiation.
18. HIV dementia or other neurologic disease that, in the judgment of the investigator, would be a contraindication to study participation.
19. Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
20. Malignancy (Not excluded from participation: Volunteer who has had malignancy excised surgically and who, in the investigator's judgment, has a reasonable assurance of sustained cure, or who is unlikely to experience recurrence of malignancy during the period of the study).
21. Current untreated or incompletely treated active tuberculosis disease or current latent tuberculosis infection (Not excluded from participation: Volunteer who has latent tuberculosis infection and is undergoing treatment, with at least one month of treatment completed)
22. Untreated or incompletely treated syphilis, gonorrhea, or chlamydia infection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-08-22 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shelly Karuna, Study Chair — HVTN Core, Fred Hutch; Katharine Bar, Study Chair — University of Pennsylvania
Locations (6):
- Instituto de Pesquisa Clinica Evandro Chagas (IPEC), FIOCRUZ, Rio de Janeiro, Brazil
- Peru (5):
  - Asociacion Civil Selva Amazonica (ACSA), Iquitos CRS, Iquitos, Maynas
  - Centro de Investigaciones Tecnológicas, Biomédicas y Medioambientales, San Marcos CRS, Callao
  - Asociacion Civil Impacta Salud y Educacion, Barranco CRS, Lima
  - Via Libra CRS, Lima
  - San Miguel CRS, Lima

RESULTS

PARTICIPANT FLOW:
Groups:
- VRC01 10mg/kg: Treatment assignment in HVTN704/HPTN 085: VRC01 10mg/kg at week (0,8,16,24,32,40,48,56,64,72)
- VRC01 30mg/kg: Treatment assignment in HVTN704/HPTN 085: VRC01 30mg/kg at week (0,8,16,24,32,40,48,56,64,72)
- Placebo: Treatment assignment in HVTN704/HPTN 085: Control for VRC01 at week (0,8,16,24,32,40,48,56,64,72)
Period: Overall Study
Arm/Group | VRC01 10mg/kg | VRC01 30mg/kg | Placebo
Started | 7 | 5 | 6
Completed | 7 | 5 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VRC01 10mg/kg | VRC01 30mg/kg | Placebo | Total
Number analyzed (Participants) | 7 | 5 | 6 | 18
Age, Continuous [Median (Full Range); unit: years] | 24 [23 to 35] | 26 [23 to 29] | 29 [24 to 44] | 27 [23 to 44]
Age, Customized [Count of Participants; unit: Participants]
  18 - 20 years | 0 | 0 | 0 | 0
  21 - 30 years | 6 | 5 | 3 | 14
  31 - 40 years | 1 | 0 | 1 | 2
  41 - 50 years | 0 | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 7 | 5 | 6 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 6 | 18
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 0 | 0 | 1 | 1
  More than one race | 0 | 0 | 0 | 0
  Other | 6 | 5 | 5 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Peru | 7 | 5 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Time to Meeting Criteria for ART Re-initiation
Description: From ART Re-Initiation Criteria form, calculated median and range of weeks of ATI meeting ART re-initiation criteria by HVTN 704/HPTN 085 treatment assignment. Note that participants with plasma ARV levels consistent with ongoing ARV use during ATI schedule are excluded
Time Frame: Measured through participant's last visit on Schedule 1 or 2, up to 6 months.
Population: Participants with plasma ARV levels consistent with ongoing ARV use during ATI schedule are excluded
Measure: Median (Full Range); unit: Weeks
Arm/Group | VRC01 10mg/kg | VRC01 30mg/kg | Placebo
Number analyzed (Participants) | 7 | 4 | 6
Weeks | 7.9 [4.6 to 20.4] | 8.9 [4.1 to 23.1] | 7.6 [2.7 to 17.9]

2. Primary Outcome: Frequency of Sustained Post-treatment HIV Control, Defined as ≥ 24 Weeks Off ART Without Meeting ART Re-initiation Criteria
Description: From ART Re-Initiation Criteria form, counts number of participants with ≥ 24 weeks of ART without meeting ART re-initiation criteria by HVTN 704/HPTN 085 treatment assignment. Note that participants with evidence of ARV use in ATI monitoring schedule are excluded from the analysis
Time Frame: Measured at week 24 of schedule 1- monitoring ATI
Population: Participants with evidence of ARV use in ATI monitoring schedule are excluded from the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | VRC01 10mg/kg | VRC01 30mg/kg | Placebo
Number analyzed (Participants) | 7 | 4 | 6
Participants | 0 | 0 | 0

3. Primary Outcome: Percentage of Participants Who Experience Adverse Events (AEs)
Description: Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017
Time Frame: Measured through participant's last study visit, up to 18 months.
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | VRC01 10mg/kg | VRC01 30mg/kg | Placebo
Number analyzed (Participants) | 7 | 5 | 6
Participants | 7 | 5 | 6

4. Primary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs)
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017 (exceptions apply).
Time Frame: Measured through participant's last study visit, up to 18 months.
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | VRC01 10mg/kg | VRC01 30mg/kg | Placebo
Number analyzed (Participants) | 7 | 5 | 6
Participants | 0 | 0 | 1

5. Primary Outcome: Number of Participants Who Discontinue ATI
Description: Tabulated by reason and HVTN 704/HPTN 085 treatment group. Note that 1. Participants with plasma ARV levels consistent with ongoing ARV use during ATI schedule are excluded; 2. Participants may meet more than one ART re-initiation criterion.
Time Frame: Measured through participant's last visit on Schedule 1 or 2, up to 6 months
Population: Note that 1. participants with plasma ARV levels consistent with ongoing ARV use during ATI schedule are excluded; 2. Participants may meet more than one ART re-initiation criterion.
Measure: Count of Participants; unit: Participants
Arm/Group | VRC01 10mg/kg | VRC01 30mg/kg | Placebo
Number analyzed (Participants) | 7 | 4 | 6
Participants
  Discontinuation of ATI due to Viral Load | 6 | 2 | 4
  Discontinuation of ATI due to CD4+ T-Cell Count | 0 | 0 | 0
  Discontinuation of ATI due to HIV-Related Syndrome | 0 | 1 | 0
  Discontinuation of ATI due to Pregnancy or Breastfeeding | 0 | 0 | 0
  Discontinuation of ATI due to Participant Request | 1 | 1 | 2
  Discontinuation of ATI due to Primary HIV Care Provider Request | 0 | 0 | 0
  Discontinuation of ATI due to CRS Clinician Decision | 1 | 0 | 0
  Discontinuation of ATI due to Other AE | 0 | 0 | 0

6. Primary Outcome: Number of Local Laboratory Values Meeting Grade 2 AE Criteria or Above
Description: The number (percentage) of participants with lab grade > 1 for alanine aminotransferase (ALT), Estimated Glomerular Filtration Rate (eFGR), Absolute Neutrophil Count, Direct Bilirubin, Hemoglobin, Platelets was summarized by arm. Only measurements with at least 1 record of grade 2 AE or above were shown in the table.
Time Frame: Measured through participant's last study visit, up to 18 months
Population: 'Overall Number of Participants Analyzed' represents participants enrolled and eligible for laboratory assessment. Participants do not have laboratory assessments if they attended the visit but laboratory specimens were not collected, missed the scheduled visit, or terminated participation in the study prior to the scheduled visit.
Measure: Count of Participants; unit: Participants
Arm/Group | VRC01 10mg/kg | VRC01 30mg/kg | Placebo
Number analyzed (Participants) | 7 | 5 | 6
Participants
  Alanine Aminotransferase (U/L) | 2 | 0 | 0
  Estimated Glomerular Filtration Rate (mL/min/1.73 m2) | 4 | 2 | 3

7. Secondary Outcome: Cumulative Incidence of Participants With First Viral Load ≥ 200 Copies/mL at Week 8, 16, and 24 of Schedule 1: Monitoring ATI
Description: The number (percentage) of participants with first viral load >= 200 by Schedule 1 week 8, 16, and 24. Participants with plasma ARV levels consistent with ongoing ARV use during ATI schedule are excluded
Time Frame: Measured for participants undergoing ATI up at week 8, 16, and 24
Population: Participants with plasma ARV levels consistent with ongoing ARV use during ATI schedule are excluded
Measure: Count of Participants; unit: Participants
Groups:
- VRC01 Pooled: Treatment assignment in HVTN704/HPTN 085: VRC01 10 mg/kg or VRC01 30 mg/kg at week (0,8,16,24,32,40,48,56,64,72)
Arm/Group | VRC01 Pooled | Placebo
Number analyzed (Participants) | 11 | 6
Participants
  Week 8 | 8 | 4
  Week 16 | 9 | 4
  Week 24 | 9 | 4

8. Secondary Outcome: Response Rate of HIV-specific CD4+ and CD8+ T-cells
Description: Measured by flow cytometry
Time Frame: Measured through participant's last study visit, on average 15 months
Reporting Status: Not Posted

9. Secondary Outcome: Magnitude of HIV-specific CD4+ and CD8+ T-cells
Description: Measured by flow cytometry
Time Frame: Measured through participant's last study visit, on average 15 months
Reporting Status: Not Posted

10. Secondary Outcome: Polyfunctionality of HIV-specific CD4+ and CD8+ T-cells
Description: Measured by flow cytometry
Time Frame: Measured through participant's last study visit, on average 15 months
Reporting Status: Not Posted

11. Secondary Outcome: Magnitude of Neutralizing Antibodies (nAb) Responses Against Autologous and Heterologous HIV Isolates
Description: Measured by TZM-bl neutralization assay
Time Frame: Measured through participant's last study visit, on average 15 months
Reporting Status: Not Posted

12. Secondary Outcome: Non-neutralizing, FcγR-mediated Antibody Effector Functions
Description: Measured by ADCC, ADCP, and virion capture
Time Frame: Measured through participant's last study visit, on average 15 months
Reporting Status: Not Posted

13. Secondary Outcome: Frequency of Dendritic Cell Activation and Maturation Markers
Description: Measured by flow cytometry or other cell phenotyping assays
Time Frame: Measured through participant's last study visit, on average 15 months
Reporting Status: Not Posted

14. Secondary Outcome: Frequency of T- and B-cell Activation and Exhaustion Markers
Description: Measured by flow cytometry or other cell phenotyping assays
Time Frame: Measured through participant's last study visit, on average 15 months
Reporting Status: Not Posted

15. Secondary Outcome: Frequency of CD4+ T Cells Carrying Intact and/or Total Pro-viral HIV DNA, Replication Competent Virus, and/or Cell-associated HIV RNA
Description: Measured by Intact Proviral DNA Assay (IPDA), Tat/rev Induced Limiting Dilution Assay (TILDA), assays detecting replication-competent virus-bearing cells, and/or measures of total proviral DNA. Cell-associated HIV-RNA may be quantitated as a measure of the transcriptionally active reservoir.
Time Frame: Measured through participant's last study visit, on average 15 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The AE reporting period is for the duration of the participant participation in this study: from study enrollment until the participant terminates. (up to 18 months)
Arm/Group | VRC01 10mg/kg | VRC01 30mg/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/5 | 1/6
Other Adverse Events (participants affected / at risk) | 7/7 | 5/5 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VRC01 10mg/kg (N=7) | VRC01 30mg/kg (N=5) | Placebo (N=6)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VRC01 10mg/kg (N=7) | VRC01 30mg/kg (N=5) | Placebo (N=6)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Acute HIV infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Acute hepatitis C (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Anal chlamydia infection (Infections and infestations) | 4 (7) | 4 (7) | 3 (6)
Furuncle (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Genitourinary tract gonococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Latent syphilis (Infections and infestations) | 4 (7) | 3 (5) | 1 (1)
Monkeypox (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (4)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal gonococcal infection (Infections and infestations) | 3 (4) | 5 (6) | 2 (2)
Parasitic gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal chlamydia infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 2 (3) | 1 (1)
Primary syphilis (Infections and infestations) | 1 (2) | 1 (1) | 2 (2)
Proctitis gonococcal (Infections and infestations) | 4 (4) | 2 (3) | 2 (2)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Secondary syphilis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urethritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urethritis chlamydial (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 2 (2) | 0 (0) | 1 (2)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 3 (4) | 1 (1) | 2 (2)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 1 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Mixed anxiety and depressive disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Balanoposthitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-03-22): https://cdn.clinicaltrials.gov/large-docs/58/NCT04801758/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-04): https://cdn.clinicaltrials.gov/large-docs/58/NCT04801758/SAP_001.pdf